CLINICAL TRIAL: NCT01599715
Title: Translating Unique Learning for Incontinence Prevention for Women Over the Age of 55
Brief Title: Translating Unique Learning for Incontinence Prevention
Acronym: TULIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Carolyn Sampselle, Carolyne K Davis Professor of Nursing, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: The TULIP Project; R01NR012011-01 (NIH)
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Weak bladder; Frequent urination; Overactive bladder; Urine leakage; Stress incontinence; Urge Incontinence; Pelvic Floor weakness; Pelvic Floor Muscle Exercises; Kegel exercises; Self-Care
MeSH Terms: conditions — Urinary Incontinence; Nocturnal Enuresis; Urinary Bladder, Overactive; Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Instructional DVD Intervention (Other): Participants randomized to this arm watched an eighteen minute bladder health instructional DVD at the conclusion of a successful baseline screening visit. This intervention occurred only once
  Interventions: Behavioral: Instructional DVD
- Bladder Health Class Intervention (Other): Participants randomized to this arm attended a two-hour bladder health instruction session that reviewed 3 primary self-care techniques that have been proven to prevent or lessen the severity of urinary incontinence. This session occurred only once 1-3 weeks subsequent to a successful baseline screening visit.
  Interventions: Behavioral: Bladder Health Class

INTERVENTIONS:
Behavioral: Instructional DVD — Participants randomized to this arm watched an eighteen minute bladder health instructional DVD at the conclusion of a successful baseline screening visit. This intervention occurred only once.
  Arms: Instructional DVD Intervention
Behavioral: Bladder Health Class — Participants randomized to this arm attended a two-hour bladder health instruction session that reviewed 3 primary self-care techniques that have been proven to prevent or lessen the severity of urinary incontinence. This session occurred only once 1-3 weeks subsequent to a successful baseline screening visit.
  Arms: Bladder Health Class Intervention

SUMMARY:
More than one in three US women suffers from the distressing, embarrassing, and often unreported problem of urinary incontinence (UI). UI severity increases with age and the financial cost exceeds $19 billion per year . The Adult Conservative Management Committee of the 2008 International Consultation on Incontinence concluded that pelvic floor muscle training (PFMT) should be offered as first line therapy to all women with stress, urge, or mixed UI; and that bladder training (BT) may be preferred to drug therapy. Conservative strategies are low risk and differ from other forms of UI management in that they do not prejudice future treatments. They also may decrease symptoms of urgency and frequency that do not entail UI, but greatly reduce the quality of life for nearly 1 in 11 US women.

DETAILED DESCRIPTION:
The study will attempt to accomplish 3 aims:

Aim 1: Compare outcomes of the two-hour BH Class with the condensed DVD version.

To accomplish this aim we will conduct a comparative effectiveness trial of 600 women 55 years and older randomized to BH Class or DVD. Women will be followed for 24 months post-intervention in order to assess long-term outcomes and sustainability.

Aim 2: Conduct an economic analysis comparing the two-hour BH Class with the DVD version. Describing the costs, quality of life, and analyzing the willingness to pay and employment/ productivity data will be the primary economic focus of this study.

Aim 3: Conduct a qualitative analysis to gain insight into elements of the intervention that contribute to sustainability.

Inclusion/Exclusion Criteria

Inclusion:

1. Female, aged 55 years or older
2. An additive sum of the frequency (question 1) and volume (question 2) items from the International Consultation on Incontinence Questionnaire-Short Form is ≤5
3. Negative for demonstrable UI on the standardized Paper Towel Test
4. Willing to undergo vaginal/pelvic examination
5. Willing and able to be compliant with visit schedule and study procedures for the study duration
6. Provide written informed consent form
7. Able to understand and read English

Exclusion:

1. Non-ambulatory (patient confined to bed or wheelchair)
2. Persistent pelvic pain (defined as daily pelvic pain)
3. History of neurologic diseases (e.g. Cerebral Vasular Accident, Parkinson's disease, Multiple sclerosis, Epilepsy, Spinal cord tumor or trauma, spina bifida, current symptomatic herniated disc)
4. Actively taking UI, OAB, or any other bladder control medication.
5. Other urinary conditions or procedures that may affect continence status (e.g. history of bladder cancer, urethral diverticula, previous augmentation cystoplasty or artificial sphincter; implanted nerve stimulators for urinary symptoms, history of sling surgery for UI or prolapse)
6. Participation in another research project that may influence the results of this trial
7. Pelvic organ prolapse protruding past the introitus upon straining
8. Absolute absence of pelvic floor muscle strength manifested by zero Brink test (Brink et al., 1994 for pressure and displacement 9
9. Evidence of UTI or hematuria - Urine dipstick positive for red blood cells will exclude the participant from enrollment in the study until a microscopic urinalysis is negative. Urine dipstick positive for leukocytes plus nitrates will exclude the participant from enrollment in the study and require further evaluation for UTI.
10. History of > 2 recurrent UTI's in the past year and no more than one UTI within 6 months
11. Post void residual > 150 cc

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 55 years or older
2. An additive sum of the frequency (question 1) and volume (question 2) items from the International Consultation on Incontinence Questionnaire-Short Form is ≤5
3. Negative for demonstrable UI on the standardized Paper Towel Test
4. Willing to undergo vaginal/pelvic examination
5. Willing and able to be compliant with visit schedule and study procedures for the study duration
6. Provide written informed consent form
7. Able to understand and read English

Exclusion Criteria:

1. Non-ambulatory (patient confined to bed or wheelchair)
2. Persistent pelvic pain (defined as daily pelvic pain)
3. History of neurologic diseases (e.g. Cerebral Vasular Accident, Parkinson's disease, Multiple sclerosis, Epilepsy, Spinal cord tumor or trauma, spina bifida, current symptomatic herniated disc)
4. Actively taking UI, OAB, or any other bladder control medication.
5. Other urinary conditions or procedures that may affect continence status (e.g. history of bladder cancer, urethral diverticula, previous augmentation cystoplasty or artificial sphincter; implanted nerve stimulators for urinary symptoms, history of sling surgery for UI or prolapse)
6. Participation in another research project that may influence the results of this trial
7. Pelvic organ prolapse protruding past the introitus upon straining
8. Absolute absence of pelvic floor muscle strength manifested by zero Brink test (Brink et al., 1994 for pressure and displacement 9
9. Evidence of UTI or hematuria - Urine dipstick positive for red blood cells will exclude the participant from enrollment in the study until a microscopic urinalysis is negative. Urine dipstick positive for leukocytes plus nitrates will exclude the participant from enrollment in the study and require further evaluation for UTI.
10. History of > 2 recurrent UTI's in the past year and no more than one UTI within 6 months
11. Post void residual > 150 cc

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2010-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Translating Unique Learning for Incontinence Prevention (TULIP) | 5 years
  Prevention study for Urinary Incontinence in women over the age of 55 who are fully continent (do not leak urine at all) or mildly continent (leak small drops of urine on occasion). This study will measure the effectiveness of 2 interventions: a bladder health instruction session or Bladder Health DVD administration.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Sampselle, PHD, RN, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan School of Nursing, Ann Arbor, Michigan
  - University of Pennsylvania Department of Urology, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Manuscript preparation for data dissemination is currently in progress.